CLINICAL TRIAL: NCT06008392
Title: INTERogating Cancer for Etiology, Prevention and Therapy Navigation (INTERCEPTioN)
Brief Title: INTERogating Cancer for Etiology, Prevention and Therapy Navigation
Acronym: INTERCEPTioN
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-008878; NCI-2024-03113 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-08-08; First posted 2023-08-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Cancer Gene Mutation; PAN Gene Mutation; Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
Keywords: Whole Exome Sequencing (WES); Whole Genome Sequencing (WGS); Genetic Testing; Genetic Counseling; Genomics
MeSH Terms: conditions — Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Biospecimen Retention: Samples With DNA — Each participant will have residual/archived tissue and a new blood (or saliva, hair follicle) sample for pan-genomic testing as per standard of care testing. Additional samples (including but not limited to tissue, bone marrow, blood, urine, stool, hair follicles, etc) may be requested/collected to be used for additional genomic and other omics studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Germline and Somatic Testing: Potential participants with a cancer diagnosis may be identified through the following sources: patients who will undergo or are currently undergoing clinical evaluation in practices such as, but not limited to, hematology-oncology, gastroenterology-hepatology, radiation-oncology and surgery. Participants will be enrolled in the study indefinitely unless a request to withdraw is made.
  Interventions: Genetic: Pan-genomic Testing
- Group B: Germline Testing Only: Potential participants with a cancer diagnosis may be identified through the following sources: patients who will undergo or are currently undergoing clinical evaluation in practices such as, but not limited to, hematology-oncology, gastroenterology-hepatology, radiation-oncology and surgery. Participants will be enrolled in the study indefinitely unless a request to withdraw is made.
  Interventions: Genetic: Pan-genomic Testing

INTERVENTIONS:
Genetic: Pan-genomic Testing — Participants will be scheduled to review the study specifics, review consent and gather medical information. Once consented, samples will be collected. When the samples are received by Exact Sciences, DNA and RNA will be extracted, and sequencing will be performed. Following pan-genomic testing, participants will receive the full report with results from their care team and results will also be added to the patient's portal. If a germline finding is identified (positive pathogenic variant) the participant will also be referred for a genetic counselor visit. All results from the germline hereditary test will be reviewed by a certified genetic counselor in addition to a review of their pedigree. To help with review of any genetic research findings, the study team may request to obtain genomic data from previous genetic testing (clinical or research based).
  Other Names: Genetic testing

SUMMARY:
This study is being done to identify markers and causes of cancer by analyzing patient's DNA (i.e., genetic material), RNA, plasma, tissues, or other samples that could be informative for patients with cancer. Cancer genetic testing is a series of tests that finds specific changes in cancer cells and normal cells in the body. Researchers may request to access these data as they explore how to better prevent, screen, or treat cancer. This study is also being done to create a biobank (library) of samples and information to learn more about treating cancer. Discovery of genetic variants in patients with cancer could result in opportunities for cancer prevention, earlier diagnosis or better therapy for cancer.

ELIGIBILITY:
Inclusion Criteria:

GROUP A: Germline and Somatic Testing

* Has Mayo Clinic medical record number
* Confirmed cancer diagnosis which is either recurrent, relapsed, refractory, metastatic, or advanced
* Participant aware of cancer diagnosis
* Able to provide informed consent
* Ability to provide blood, saliva, bone marrow aspirate or hair follicle sample
* Ability to provide archived tissue, Note: if tissue unavailable participant may still enroll onto the study for the germline collection, or vice versa, if germline has already been completed may still enroll for somatic tissue testing.

GROUP B: Germline testing only:

* Has Mayo Clinic medical record number
* Confirmed cancer diagnosis
* Participant aware of cancer diagnosis
* Able to provide informed consent
* Ability to provide blood, saliva, or hair follicle sample

Exclusion Criteria:

Note: Women who are pregnant or planning to become pregnant can take part in this study.

GROUP A: Germline and Somatic testing

* Individuals who have situations that would limit compliance with the study requirements
* Institutionalized (i.e. Federal Medical Prison)
* Prior germline genetic testing with a 100+ multi-gene panel within the last 1 year of enrollment, AND/OR
* Prior somatic tissue (250+ gene) testing within the prior 3 months of enrollment

GROUP B: Germline testing only

* Individuals who have situations that would limit compliance with the study requirements
* Institutionalized (i.e. Federal Medical Prison)
* Prior germline genetic testing with a 100+ multi-gene panel within the last 1 year of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants identified internally to Mayo Clinic will be enrolled. The Mayo Clinic study team and/or subspecialty teams will identify participants that fulfill enrollment criteria. Only individuals with a confirmed cancer diagnosis who know they have cancer will be asked to participate. Group B will enroll patients who do not meet NCCN and CMS guidelines for somatic tissue testing and/or whom have had somatic tissue testing, but not germline testing previously.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2033-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Genomic sequencing of tumor tissue and blood | Baseline; 50 years
  Genomic sequencing of tumor tissue and blood will be performed to determine genomic alterations in germline and somatic cancer-related genes (SNVs, indels, CNVs from DNA and fusions from RNA) to allow the ordering hematologist/oncologist/provider to determine optimal therapy and clinical trial prospective. Researchers across the field of genomic sequencing report findings about new variations in scientific publications and collect it in databases every day. Consequently, any patient's variant of uncertain significance (VUS) result could be reclassified by emerging findings, turning previously unresolved tests into diagnostic answers. Our Translational Omics Program has a system to re-analyze a patient's exome/genome data against these new genetic findings-reviewing data and comparing it with emerging clinical genetic data to facilitate diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Jewel J. Samadder, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials